CLINICAL TRIAL: NCT01041560
Title: Muscle Tone Changes in Acute Stroke According to Brain Injury in Relation to Changes in Functioning
Brief Title: Muscle Tone Changes in Acute Stroke According to Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jyväskylä Central Hospital (Other)
Collaborators: Eurostars (Other)
Responsible Party: Ylinen Jari, MD, PhD, Jyväskylä Central Hospital
Other Study IDs: KSKS2
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2009-12-31 (Estimated); Status verified 2009-12

CONDITIONS: Stroke
Keywords: Stroke; Tone; Strength
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stoke: Hemiplegia with unilateral changes in tone and muscle strength

SUMMARY:
The purpose of the study is to examine connections between muscle tones, strength and function after stroke.

DETAILED DESCRIPTION:
Measurements are intended to repeat every two days in acute phase to discover possible changes in tone and strength in arm and leg muscles.

ELIGIBILITY:
Inclusion Criteria:

* unilateral decline in the arm or leg muscle strength

Exclusion Criteria:

* unwilling to take part on the trial
* not conscious
* no differences between muscle strength on the right and left side

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients in Middle-Finland Central hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Muscle tone | Immediately after stroke, during the first week in hospital every other day, and then once a week before discharging from hospital

SECONDARY OUTCOMES:
Muscle strength | Immediately after stroke, during the first week in hospital every other day, and then once a week before discharging from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jari Ylinen, MD, PhD, Study Director — Senior physician
Locations (1):
- Central Finland Health Care District, Jyväskylä, Finland